CLINICAL TRIAL: NCT05984303
Title: Treatment of Decompensated Cirrhosis Using Human Umbilical Cord-derived Mesenchymal Stem Cells: A Phase 1, Multiple Administration, Dose-escalasion Trial (MSC-DLC-1b)
Brief Title: Human Umbilical Cord-derived Mesenchymal Stem Cells for Decompensated Cirrhosis (MSC-DLC-1b)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Wuhan Optics Valley Zhongyuan Pharmaceutical Co., Ltd., Hubei, China (Unknown)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-DLC-1b
Record Dates: First submitted 2023-07-28; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Cord-derived Mesenchymal Stem Cells (Experimental): Standard of care (SOC) plus a multiple administration and dose-escalasion with 2 cohorts with 3 subjects/cohort who receive doses of 1 and 2 ×10E8 cells. Each person received 3 infusions, 1 week apart, Proceed from lower dose to higher dose if no safety concerns for each cohort.
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord-derived Mesenchymal Stem Cells — Human Umbilical Cord-derived Mesenchymal Stem Cells will be administered intravenously.

SUMMARY:
This clinical trial is a Phase 1, multiple administration, dose-escalasion clinical trial of human umbilical cord-derived mesenchymal stem cells for the treatment of decompensated cirrhosis. The primary objective of this study is to assess the safety of intravenous infusion of human umbilical cord-derived mesenchymal stem cells in patients with decompensated cirrhosis.

DETAILED DESCRIPTION:
Decompensated cirrhosis has a high overall mortality rate. There is unmet need for safe and alternative therapeutic potions. This clinical trial is a Phase 1, multiple administration, dose-escalasion clinical trial of human umbilical cord-derived mesenchymal stem cells for the treatment of decompensated cirrhosis. The primary objective of this study is to assess the safety of intravenous infusion of human umbilical cord-derived mesenchymal stem cells in patients with decompensated cirrhosis.In order to illustrate the safety and effectiveness of human umbilical cord-derived mesenchymal stem cells and the patient's dose tolerance to human umbilical cord-derived mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Aged 18 to 75 years (including 18 and 75 years), male or female;
3. Patients diagnosed with decompensated liver cirrhosis based on clinical findings, laboratory tests, imaging findings and/or representative pathological findings (decompensated liver cirrhosis is defined as the occurrence of at least one serious complication, including esophageal and gastric varices bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis and other serious complications);
4. Child-Turcotte-Pugh (CTP) score 7 to 12 points.

Exclusion Criteria:

1. Hepatitis B virus (HBV) DNA ≥ detection limit at the time of screening, or patients with hepatitis B virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HBV for less than 12 months.
2. Hepatitis C virus (HCV) RNA ≥ detection limit at the time of screening, or patients with hepatitis C virus-related decompensated liver cirrhosis not more than 12 months on antiviral therapy.
3. Patients under treatment with corticosteroids for autoimmune hepatitis for less than 6 months.
4. Trans-jugular intrahepatic portosystemic shunts (TIPS) insertion within 6 months prior to study inclusion.
5. Active drinkers with alcohol-related decompensated cirrhosis are unwilling to stop alcohol abuse after inclusion.
6. Patients with biliary obstruction, or portal patients with vein spongiosis.
7. Patients are known with other malignancies within 5 years prior to the signing of ICF, except have had curative therapy of Basal Cell Cancer, Squamous Cell Carcinoma and/or radical resection of Carcinoma in Situ.

   Known to have had other malignancies within 5 years prior to signing the informed consent, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ with curable resection.
8. Patients with history of organ transplantation.
9. Patients with severe heart, lung, kidney and blood system diseases.
10. Patients with drug abuse, drug dependence and patients who receive methadone treatment or with psychosis.
11. Patients with history of immunodeficiency disease, including a positive test result for human immunodeficiency virus (HIV) antibodies, or other acquired or congenital immunodeficiency diseases;
12. Pregnant or lactating female. Fertile patients who were unable or unwilling to use effective non-pharmaceutical contraception during the trial and within 6 months after the end of the trial.
13. Patients who had cardiovascular and cerebrovascular events (such as Unstable Angina, Brain Hemorrhage, severe Ischemic Infarction) within 3 months before the first dose；Patients who had Myocardial Infarct or a clinically significant Arrhythmia/Conduction Abnormalities within 12 months before the first dose.
14. Patients with hypersensitivity (allergic to more than two foods or drugs) or with a history of severe allergy, or patients with Severe allergy to a known experimental drug or to any excipient.
15. Patients previously received stem cell therapy or are intolerance to cell therapy;
16. Participants in other clinical trials within the last 3 months.
17. Any other clinical condition which the investigator considers would make the patient unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | from baseline to 28th day
incidence of dose-limiting toxicity-related adverse events | from baseline to 28th day
maximum tolerated dose | from baseline to 28th day
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 28th day | at 28th day
  The Model for End-stage Liver Disease (MELD) is a scoring system that evaluates the liver function reserve and prognosis of patients with chronic liver disease by creatinine, international normalized ratio (INR), and bilirubin-conjugated cirrhosis etiology.
  The MELD score is calculated by the formula: R = 9.6 × ln (creatinine mg/dl) + 3.8 × ln (bilirubin mg/dl) + 11.2 × ln (INR) + 6.4 × etiology, and the results are taken as integers. ( 0 for cholestatic and alcoholic cirrhosis and 1 for other causes of cirrhosis such as viruses).

SECONDARY OUTCOMES:
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 3 days, 7days, 14 days, 21 days, 1 month, 2 months, 3 months, 6 months, 12 months, 18 months, and 24 months | 3 days, 7days, 14 days, 21 days, 1 month, 2 months, 3 months, 6 months, 12 months, 18 months, and 24 months
Incidence of each complication associated with decompensated cirrhosis | up to 24 months
liver transplant-free survival | up to 24 months
Incidence of liver failure | up to 24 months
plasma albumin (ALB) | up to 24 months
plasma prealbumin (PALB) | up to 24 months
total bilirubin (TBIL) | up to 24 months
serum cholinesterase (CHE) | up to 24 months
prothrombin time (PT) | up to 24 months
  Prothrombin time (PT) is a blood test that measures the time it takes for plasma to clot, to check for bleeding problems, or to check whether medicine to prevent blood clots is working.
Child-Turcotte-Pugh (CTP) score | up to 24 months
  Child-Turcotte-Pugh (CTP) score is a scoring system that evaluates the liver function.
  Maximum is 15, minimum is 5. Higher scores mean a worse outcome.
EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D) | up to 24 months
  Quality of life assessment. Maximum is 5, minimum is 1. Lower scores mean a better outcome.
Incidence of liver cancer | up to 24 months
ChronicLiver Disease Questionnaire (CLDQ) | up to 24 months
  Quality of life assessment. The Chronic Liver Disease Questionnaire (CLDQ) was developed as an evaluative instrument to measure longitudinal change in health status within individuals with chronic liver disease. In addition to measuring both physical and mental health, the instrument was designed to be a disease-specific tool for assessing areas of function important to patients with chronic liver disease. Maximum is 7, minimum is 1. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, PhD, Study Chair — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.

REFERENCES:
- [Derived] Shi L, Zhang Z, Mei S, Wang Z, Xu Z, Yao W, Liu L, Yuan M, Pan Y, Zhu K, Liu K, Meng F, Sun J, Liu W, Xie X, Dong T, Huang L, Meng F, Fu JL, Li Y, Zhang C, Fan X, Shi M, Zhang Y, Li Y, Xie WF, Zhang P, Wang FS. Dose-escalation studies of mesenchymal stromal cell therapy for decompensated liver cirrhosis: phase Ia/Ib results and immune modulation insights. Signal Transduct Target Ther. 2025 Jul 29;10(1):238. doi: 10.1038/s41392-025-02318-4. PMID 40721581